CLINICAL TRIAL: NCT01727037
Title: A Feasibility and Safety Study of Bronchoscopic Intrabullous Autologous Blood Instillation for the Treatment of Severe Bullous Emphysema (BIABI Study)
Brief Title: Bronchoscopic Intrabullous Autologous Blood Instillation (BIABI) for Emphysema
Acronym: BIABI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIABI v1
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Bullous Emphysema
Keywords: Emphysema; Chronic obstructive pulmonary disease; COPD; Bulla; Interventional bronchoscopy; Lung volume reduction
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Blister

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIABI arm (Experimental): Patients will undergo intrabullous autologous blood instillation
  Interventions: Procedure: Bronchoscopic intrabullous autologous blood instillation

INTERVENTIONS:
Procedure: Bronchoscopic intrabullous autologous blood instillation
  Other Names: BIABI

SUMMARY:
Patients with large bullae (large empty air sacs in the lung) may benefit from bullectomy (surgery to resect these bullae), however this is a major surgery with significant potential morbidity and long hospital stays. Many patients are not well enough to have this surgery, or may not wish to have it. A less invasive means of attempting to shrink the size of the bullae is to directly inject the patients' own blood into the bullae (we believe that this can lead to an inflammatory reaction leading to gradual scarring and volume loss). This can be performed bronchoscopically in a 20-30 minute procedure using conscious sedation (avoiding general anaesthesia).

The aim of this study is to assess the effects on lung function, quality of life measures, functional measures and CT measured lung volumes of bronchoscopic intrabullous blood instillation in patients with bullous emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Age > 35 years
* Large bulla on CT scan where bullectomy is contraindicated or is actively avoided.
* Hyperinflation - TLC ≥100% predicted, RV ≥150% predicted
* Exertional breathlessness (mMRC >0)
* Optimum COPD treatment for at least 6 weeks
* No COPD exacerbation for at least 6 weeks
* Fewer than 3 admissions for infective exacerbations in the preceding 12 months
* Written informed consent

Exclusion Criteria:

* Inability to obtain informed consent
* Co-morbidities that would render bronchoscopy or sedation unsafe.
* Anaemia or other reasons precluding venesection.
* Clinically significant bronchiectasis
* Arrhythmia or cardiovascular disease that poses a risk during procedure
* Lung nodule requiring further investigation or treatment
* Subject taking clopidogrel, warfarin, or other anticoagulants and unable to abstain for 5 days pre-procedure

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Change in the Residual Volume (RV) following treatment | 6 months

SECONDARY OUTCOMES:
Change in TLC 6 months following treatment | 6 months
Change in RV/TLC ratio 6 months following treatment | 6 months
Changes in FEV1 and FVC 6 months following treatment | 6 months
Change in the intrathoracic gas volume 6 months following treatment | 6 months
Change in DLCOc 6 months following treatment | 6 months
Change in the SGRQ score 6 months following treatment | 6 months
Change in the mMRC score 6 months following treatment | 6 months
Change in the 6MWD 6 months following treatment | 6 months
Change in CT measured lung volumes 6 months following treatment | 6 months
Adverse events | 6 monhts

CONTACTS AND LOCATIONS:
Overall Officials: Pallav L Shah, MD FRCP, Principal Investigator — Royal Brompton and Chelsea and Westminster Hospitals
Locations (3):
- United Kingdom (3):
  - Kings Mill Hospital, Sherwood Forest Hospitals NHS Trust, Mansfield, Nottinghamshire,
  - The Royal Brompton and Harefield NHS Trust, London
  - Chelsea and Westminster Hospital NHS Foundation trust, London